CLINICAL TRIAL: NCT00759889
Title: Obtaining and Storing Standard of Care Wound Biopsies for Immediate or Future Wound Related Scientific Study
Brief Title: Obtaining and Storing Standard of Care Wound Biopsies for Immediate or Future Wound-Related Scientific Study
Status: Completed | Type: Observational
Sponsor: Southwest Regional Wound Care Center (Other)
Responsible Party: Principal Investigator, Randall Wolcott, Prinicipal Investigator, Southwest Regional Wound Care Center
Other Study IDs: 56-RW-005
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Diabetic Foot; Leg Ulcer; Decubitus Ulcer
Keywords: venous leg ulcer
MeSH Terms: conditions — Diabetic Foot; Leg Ulcer; Pressure Ulcer; Varicose Ulcer

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Wound edge biopsies that are obtained through standard of care protocols will be subjected to additional microscopic and molecular analyses following the completion of standard medical assessment.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- wound biopsy: diabetic foot,venous leg ulcer, decubitus ulcer

SUMMARY:
The objective of this study protocol is to use wound biopsies that have been obtained during standard of care management for further scientific evaluation after standard evaluation by a pathologist. Further imaging and molecular analyses would closely evaluate the presence, architecture, and interaction of wound biofilm and human host tissues.

DETAILED DESCRIPTION:
The criteria for considering a wound biopsy in a given patient are a chronic wound (venous leg ulcer, diabetic foot ulcer, decubitus ulcer) that has been present for over two (2) months and has failed to progress towards healing (less than 20% decrease in size over 2-week period of time). Also any suspicious wound in which cancer is strongly considered on a clinical basis should be biopsied immediately without any arbitrary timeline being imposed.

ELIGIBILITY:
Inclusion Criteria:

* The subject must have a wound, which requires a biopsy for at least one of the following reasons:

  * The wound is clinically suspicious (raised fibrotic edges, patchy discoloration of the edges, "invasive appearance", or an appearance substantially different from normal chronic wound appearance).
  * The wound has been present for over 3 months that has been under standard of care management for at least 1 month and shows no progression towards healing. No progression towards healing is defined as less than 20% reduction in the size of the wound over a 2-week period of time.
* The subject must be at least 18 years of age.
* The ulcer to be biopsied must be greater than 3 centimeters in area.

Exclusion Criteria:

* Unacceptable risk of bleeding as determined by the investigator.
* Medical or emotional risk associated with the potential biopsy that outweighs the risk of not taking a biopsy as determined by the investigator.

  * Note: Vulnerable populations will not be excluded from the study as they are over represented in the chronic wound population, but care will be taken to explain the study to family members and caretakers and other stakeholders in the subject's care, so that concerned parties are in agreement as to the subject's enrollment in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Wound edge biopsies that are obtained through standard of care protocols will be subjected to additional microscopic and molecular analyses following the completion of standard medical assessment.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2007-03 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
To analyze and image wounds using microscopy and molecular techniques | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Randall Wolcott, MD, Principal Investigator — Southwest Regional Wound Care Center
Locations (1):
- Southwest Regional Wound Care Center, Lubbock, Texas, United States